CLINICAL TRIAL: NCT00544180
Title: Record on Satisfaction of Patients With Actonel 35 mg Once a Week
Brief Title: ROSPA - Record on Satisfaction of Patients With Actonel 35 mg Once a Week
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated due to lack of compliance with GCP regulations.
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RISED_L_01686
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Risedronate

SUMMARY:
To determine the satisfaction of subject with Actonel 35 mg Once a Week in the treatment of post-menopausal osteoporosis. Open, non-controlled, multi-center study.

ELIGIBILITY:
Inclusion criteria :

* Postmenopausal ambulatory women
* Established osteoporosis

Exclusion criteria:

* History of cancer: basal cell or squamous cell carcinoma-documented 6-month remission,
* Diagnosis of hypocalcemia, hyperparathyroidism, hyperthyroidism

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction and compliance | During all the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Chantelot, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Netanya, Israel